CLINICAL TRIAL: NCT06712407
Title: An Open-label Study to Assess the Efficacy and Safety of Extended TARPEYO® (Delayed-release Budesonide Capsules) Treatment in Adult Patients With Primary IgA Nephropathy Who Have Completed 9 Months of TARPEYO® 16 mg Once Daily Treatment in Real-world Clinical Practice
Brief Title: Efficacy and Safety of Extended TARPEYO® Treatment Beyond 9 Months in Adult Patients With Primary IgA Nephropathy
Acronym: NefXtend
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Nef-403
Record Dates: First submitted 2024-11-20; First posted 2024-12-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: IgA Nephropathy
Keywords: TARPEYO®; IgAN; urine protein-to-creatinine; ESRD; Nefecon
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Failure, Chronic | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: There are 2 treatment periods with the study drug:
  * TARPEYO® 16 mg (4 capsules) once a day for 6 months
  * TARPEYO® 8 mg (2 capsules) once a day for 9 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 16 mg QD then 8 mg QD (Experimental): 6-months of TARPEYO® 16 mg QD then 9-month Treatment Period with TARPEYO® 8 mg QD and TARPEYO®4 mg QD for 2 weeks for tapering.
  Interventions: Drug: TARPEYO®

INTERVENTIONS:
Drug: TARPEYO® — 6-months of TARPEYO® 16 mg QD then 9-month Treatment Period with TARPEYO® 8 mg QD and TARPEYO®4 mg QD for 2 weeks for tapering.
  Other Names: delayed-release budesonide capsules

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of extended TARPEYO® (delayed-release budesonide capsules) treatment in adult patients with primary IgA nephropathy who have completed 9 months of TARPEYO® 16 mg once daily treatment in real-world clinical practice. The main question it aims to answer is:

Is there a treatment benefit of TARPEYO® 16 mg QD extended use?

Participants will

* take part in this study for about 19 months
* Have urine tests done
* Have blood samples taken
* Have physical examinations done

DETAILED DESCRIPTION:
This clinical trial will investigate the efficacy and safety of TARPEYO® treatment extended for an additional 15 months in adult IgAN participants who have completed their initial, single 9-month TARPEYO® 16 mg QD commercial treatment regimen. Participants with residual proteinuria will be eligible for enrollment. The Treatment Period will consist of a 6-month Treatment Period with TARPEYO® 16 mg QD, followed by a 9-month Treatment Period with TARPEYO® 8 mg QD. This will be followed by a 3-month Follow-up Period, which includes the first 2 weeks of Tapering Period with TARPEYO® 4 mg QD.

The overall aim of the extended treatment is to improve and maintain the treatment effect with reduced proteinuria and protection of kidney function over a total of 2 years of TARPEYO® treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed IgAN with biopsy verification
2. Female or male participants ≥18 years of age
3. Completion of a single, initial 9 months of treatment with TARPEYO® 16 mg QD at the Baseline visit
4. Access to retrospective local laboratory assessment data on UPCR and serum creatinine. Available retrospective data should include at least 1 assessment timepoint within 3 months prior to the first dose of TARPEYO® commercial treatment.
5. On stable treatment with renin-angiotensin system (RAS) inhibitor therapy or sparsentan for at least 8 weeks prior to the Baseline visit. A stable dose is defined as a dose within 25% of the dose at Baseline.
6. If on current treatment with sodium-glucose cotransporter-2 (SGLT2) inhibitor, the treatment should have been stable for at least 8 weeks prior to the Baseline visit. A stable dose is defined as a dose within 25% of the dose at Baseline.

Exclusion Criteria:

1. Participants who have been treated with systemic immunosuppressive medications including glucocorticosteroids (GCS) other than TARPEYO® during the TARPEYO® commercial treatment period. Topical or inhalation products containing GCS or immunosuppressants are allowed.
2. Presence of other glomerulopathies (e.g., C3 glomerulopathy, diabetes nephropathy and/or hypertensive nephropathy).
3. Presence of nephrotic syndrome (i.e., proteinuria >3.5 g per day and serum albumin <3.0 g/dL, with or without edema).
4. Presence of medical condition excluding continued TARPEYO® treatment, as assessed by the Investigator.
5. On current or planned dialysis.
6. Undergone kidney transplant.
7. Poorly controlled diabetes mellitus or hypertension, as assessed by the Investigator.
8. Participants with known osteoporosis in the medium- or high-risk category according to the 2010 American College of Rheumatology recommendations.
9. Any medical or social circumstance making trial participation and/or TARPEYO® treatment unsuitable, as assessed by the Investigator.
10. Participants with clinically significant infections that put the participant at risk, at the discretion of the Investigator.
11. Participants unwilling or unable to meet the requirements of the protocol.
12. Intake of another investigational drug during trial, or during the preceding 9-monthcommercial TARPEYO® treatment period.
13. Females who are pregnant, breastfeeding, or plan to become pregnant in the trial period.
14. Participants taking potent inhibitors of cytochrome P450 (CYP) 3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Ratio of Urine Protein to Creatine Ratio (UPCR) at 6 months compared to Baseline | 6 months
  The outcome is measured as UPCR (based on 24-hour urine collection) at 6 months following the first dose of TARPEYO® trial treatment compared to study Baseline. Ratio being UPCR at 6 months in g/gram divided with UPCR at Baseline in g/gram.

SECONDARY OUTCOMES:
Ratio of Urine Protein to Creatine Ratio (UPCR) at 15 months compared to Baseline | 15 months
  The outcome is measured as UPCR (based on 24-hour urine collection) at 15 months following the first dose of TARPEYO® trial treatment compared to study Baseline. Ratio being UPCR at 15 months in g/gram divided with UPCR at Baseline in g/gram.
Ratio of Urine Protein to Creatine Ratio (UPCR) at 6 months compared to prior to start of TARPEYO® commercial treatment (i.e., comparison with retrospective local laboratory data from medical records as available) | 18 months
  Ratio of UPCR (based on 24-hour urine collection) at 6 months compared to prior to start of TARPEYO® commercial treatment (i.e., comparison with retrospective local laboratory data from medical records as available). Retrospective data will be collected up to 3 months prior to start of commercial treatment and during the duration of the commercial treatment. Ratio being UPCR at 6 months in g/gram divided with UPCR prior to commercial treatment in g/gram
Ratio of Urine Protein to Creatine Ratio (UPCR) at 15 months compared to prior to start of TARPEYO® commercial treatment (i.e., comparison with retrospective local laboratory data from medical records as available) | 27 months
  Ratio of UPCR (based on 24-hour urine collection) at 15 months compared to prior to start of TARPEYO® commercial treatment (i.e., comparison with retrospective local laboratory data from medical records as available). Retrospective data will be collected up to 3 months prior to start of commercial treatment and during the duration of the commercial treatment. Ratio being UPCR at 6 months in g/gram divided with UPCR prior to commercial treatment in g/gram
Ratio of estimated glomerular filtration rate (eGFR) at 6 months compared to Baseline | 6 months
  The outcome is measured as ratio of eGFR in mL/min/1.73 m2 (calculated using the CKD-EPI formula) at 6 months following the first dose of TARPEYO® trial treatment compared to study baseline.
Ratio of estimated glomerular filtration rate (eGFR) at 15 months compared to Baseline | 15 months
  The outcome is measured as ratio of eGFR in mL/min/1.73 m2 (calculated using the CKD-EPI formula) at 15 months following the first dose of TARPEYO® trial treatment compared to study baseline.
Ratio of estimated glomerular filtration rate (eGFR) at 6 months compared to start of TARPEYO® commercial treatment (i.e., comparison with retrospective local laboratory data from medical records as available) | 18 months
  The outcome is measured as ratio of eGFR in mL/min/1.73 m2 (calculated using the CKD-EPI formula) at 6 months following the first dose of TARPEYO® trial treatment compared to start of commercial treatment. Retrospective data will be collected up to 3 months prior to start of commercial treatment and during the duration of the commercial treatment.
Ratio of estimated glomerular filtration rate (eGFR) at 15 months compared to start of TARPEYO® commercial treatment (i.e., comparison with retrospective local laboratory data from medical records as available) | 27 months
  The outcome is measured as ratio of eGFR in mL/min/1.73 m2 (calculated using the CKD-EPI formula) at 15 months following the first dose of TARPEYO® trial treatment compared to start of commercial treatment. Retrospective data will be collected up to 3 months prior to start of commercial treatment and during the duration of the commercial treatment.
Ratio of 24-hour urine proteinuria at 6 months compared to Baseline | 6 months
  The outcome is measured as proteinurea (based on 24-hour urine collection) at 6 months following the first dose of TARPEYO® trial treatment compared to study Baseline. Ratio being proteinurea at 6 months in g/day divided with proteinurea at Baseline in g/day.
Ratio of 24-hour urine proteinuria at 15 months compared to Baseline | 15 months
  The outcome is measured as proteinurea (based on 24-hour urine collection) at 6 months following the first dose of TARPEYO® trial treatment compared to study Baseline. Ratio being proteinurea at 15 months in g/day divided with proteinurea at Baseline in g/day.
Proportion of participants with microhematuria at 6 months | 6 months
  Number of participants with microhematuria at 6 months divided by total number of participants.
Proportion of participants with microhematuria at 15 months | 15 months
  Number of participants with microhematuria at 15 months divided by total number of participants.
To evaluate the safety (SAEs and AEs) of extended TARPEYO® treatment | 19 months
  SAEs and AEs will be evaluated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Krassimir Mitchev, Study Director — Calliditas Therapeutics
Locations (38):
- United States (37):
  - Univ of Alabama/Birmingham, Birmingham, Alabama
  - Arizona Kidney Disease & Hypertension Centers (AKDHC), Glendale, Arizona
  - The Medical Research Group, Inc., Fresno, California
  - UCI Health-UCI Medical Center, Orange, California
  - Loma Linda University, San Bernardino, California
  - UCSF Health-UCSF Medical Center-Parnassus - Nephrology and Hypertension Faculty Practice, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Hospital (UCH) - Kidney Disease and Hypertension Clinic - Anschutz Medical Campus Location, Aurora, Colorado
  - Yale University Nephrology Clinical Trials Program, New Haven, Connecticut
  - Florida Kidney Physicians, Boca Raton, Florida
  - Central Florida Kidney Specialists, Orlando, Florida
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Cobb Nephrology Hypertension Associates, PC, Austell, Georgia
  - Georgia Nephrology, Lawrenceville, Georgia
  - University of Louisville, Louisville, Kentucky
  - Ochsner Health, New Orleans, New Orleans, Louisiana
  - University of Maryland Division of Nephrology, Baltimore, Maryland
  - Boston Medical Center; Boston University Chobanian & Avedisian School of Medicine, Boston, Massachusetts
  - University of Minnesota Health Fairview, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Renal Medical Associates, Albuquerque, New Mexico
  - New York Nephrology Vasculitis and Glomerular Center, Clifton Park, New York
  - Chinatown Kidney Care, PLLC, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - North Carolina Nephrology, P.A, Raleigh, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University (OHSU) - Nephrology and Hypertension Clinic, Portland, Oregon
  - University of Pennsylvania Philadelphia, Philadelphia, Pennsylvania
  - Dallas Renal Group, Dallas, Texas
  - MedResearch Inc, El Paso, Texas
  - The University of Texas Medical Branch UTMB, Galveston, Texas
  - Memorial Hermann Houston, Houston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - The Kidney Institute/Houston, Houston, Texas
  - Dallas Nephrology Associates McKinney, McKinney, Texas
  - Permian Basin Kidney Center, Odessa, Texas
- Advanced Renal Care Institute, Mayagüez, Puerto Rico

IPD SHARING:
Plan to Share IPD: No